CLINICAL TRIAL: NCT00095030
Title: A Phase 3, Randomized, Three-Arm, Double-blind, Active Controlled, Parallel Group, Multicenter Trial to Evaluate the Safety and Efficacy of Muraglitazar in Combination With Metformin Compared to Glimepiride in Combination With Metformin in Subjects Wtih Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Therapy Alone
Brief Title: Study Comparing Muraglitazar With Glimepiride in Type 2 Diabetics Who Are Not Controlled With Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-048
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — muraglitazar

INTERVENTIONS:
Drug: muraglitazar

SUMMARY:
The purpose of this clinical research study is to learn whether a muraglitazar-metformin combination is at least as effective as a glimepiride-metformin combination to treat type 2 diabetics who are not sufficiently controlled with metformin alone. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 2 diabetes receiving treatment with at least 1,500 mg but not greater than 3000 mg of stable metformin therapy for at least 6 weeks prior to screening
* HbA1c >or = 7% and < or = 10%
* Fasting c-peptide > or = 1.0 umol
* Body Mass Index < or = 41 kg/m2
* Mean serum triglycerides < or = 600 mg/dl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1752
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in baseline HbA1c after 52 weeks

SECONDARY OUTCOMES:
Change in lipids after 52 weeks; safety and efficacy when administered with metformin after 52 weeks

CONTACTS AND LOCATIONS:
Locations (206):
- United States (108):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Fayetteville, Arkansas
  - Local Institution, Jonesboro, Arkansas
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Sherwood, Arkansas
  - Local Institution, Artesia, California
  - Local Institution, Bellflower, California
  - Local Institution, Cudahy, California
  - Local Institution, Encino, California
  - Local Institution, Fresno, California
  - Local Institution, Huntington Beach, California
  - Local Institution, Long Beach, California
  - Local Institution, Mission Viejo, California
  - Local Institution, Moreno Valley, California
  - Local Institution, Northridge, California
  - Local Institution, Paramount, California
  - Local Institution, Pasadena, California
  - Local Institution, Roseville, California
  - Local Institution, Spring Valley, California
  - Local Institution, Torrance, California
  - Local Institution, Walnut Creek, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Clearwater, Florida
  - Local Institution, DeLand, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Kissimmee, Florida
  - Local Institution, Longwood, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, Ormond Beach, Florida
  - Local Institution, Palm Harbor, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Saint Augustine, Florida
  - Local Institution, Saint Cloud, Florida
  - Local Institution, Tallahassee, Florida
  - Local Institution, Winter Park, Florida
  - Local Institution, Blue Ridge, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Chicago Heights, Illinois
  - Local Institution, Elkhart, Indiana
  - Local Institution, Slidell, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Towson, Maryland
  - Local Institution, Swansea, Massachusetts
  - Local Institution, Rolling Fork, Mississippi
  - Local Institution, Chesterfield, Missouri
  - Local Institution, Excelsior Springs, Missouri
  - Local Institution, Florissant, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, Springfield, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Toms River, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, West Seneca, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Morehead City, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Sparta, North Carolina
  - Local Institution, Statesville, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Newark, Ohio
  - Local Institution, Youngstown, Ohio
  - Local Institution, Zanesville, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Eugene, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Camp Hill, Pennsylvania
  - Local Institution, Fleetwood, Pennsylvania
  - Local Institution, Norristown, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, West Chester, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Greer, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Bristol, Tennessee
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Bryan, Texas
  - Local Institution, Corpus Christi, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Midland, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Richmond, Virginia
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Olympia, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Tacoma, Washington
  - Local Institution, Wenatchee, Washington
- Argentina (8):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Chacabuco, Buenos Aires
  - Local Institution, El Palomar, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, Buenos Aires
  - Local Institution, Córdoba
  - Local Institution, Mendoza
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Brazil (8):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Brasília, Federal District
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (29):
  - Local Institution, Calgary, Alberta
  - Local Institution, Red Deer, Alberta
  - Local Institution, Delta, British Columbia
  - Local Institution, Kelowna, British Columbia
  - Local Institution, North Vancouver, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, London, Ontario
  - Local Institution, North York, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Peterborough, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Woodstock, Ontario
  - Local Institution, York, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Chicoutimi, Quebec
  - Local Institution, Drummondville, Quebec
  - Local Institution, Fleurimont, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Germany (11):
  - Local Institution, Künzing
  - Local Institution, Magdeburg
  - Local Institution, München
  - Local Institution, Nuremberg
  - Local Institution, Rodgau
  - Local Institution, Rotenburg / Fulda
  - Local Institution, Schönebeck
  - Local Institution, Ulm
  - Local Institution, Viernheim
  - Local Institution, Vs-Schwenningen
  - Local Institution, Witten
- Hong Kong (3):
  - Local Institution, Chai Wan
  - Local Institution, Hong Kong
  - Local Institution, Shatin
- Mexico (8):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
  - Local Institution, Chihuahua City
  - Local Institution, Durango
- Peru (2):
  - Local Institution, Arequipa
  - Local Institution, Lima
- Philippines (5):
  - Local Institution, Cavite
  - Local Institution, Cebu
  - Local Institution, Manila
  - Local Institution, Pasig
  - Local Institution, Quezon
- Poland (7):
  - Local Institution, Gorzów Wielkopolski
  - Local Institution, Krakow
  - Local Institution, Mroków
  - Local Institution, Stalowa Wola
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Zabrze
- Puerto Rico (4):
  - Local Institution, Carolina
  - Local Institution, Ponce
  - Local Institution, Rio Piedras
  - Local Institution, San Juan
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
- Local Institution, Baden, Switzerland
- Taiwan (4):
  - Local Institution, Changhua
  - Local Institution, Hualien City
  - Local Institution, Taichung
  - Local Institution, Tainan
- Local Institution, Bangkok, Thailand

REFERENCES:
- [Derived] Rubin CJ, Ledeine JM, Fiedorek FT. Improvement of glycaemic and lipid profiles with muraglitazar plus metformin in patients with type 2 diabetes: an active-control trial with glimepiride. Diab Vasc Dis Res. 2008 Sep;5(3):168-76. doi: 10.3132/dvdr.2008.028. PMID 18777489